CLINICAL TRIAL: NCT04798651
Title: Pathogenicity of B and CD4 T Cell Subsets in Multiple Sclerosis
Acronym: T4MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2020/71
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: Autoimmune Diseases of the Nervous System; Multiple sclerosis; clinically isolated syndrome; lymphoid cells; CD4 T cells; B cells
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases of the Nervous System | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with multiple sclerosis or clinically isolated syndrome (Experimental): subjects with MS defined by 2010 revised McDonald criteria or presenting a clinical isolated syndrome
  Interventions: Biological: blood sample; Biological: cerebro-spinal fluid

INTERVENTIONS:
Biological: blood sample — 28 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Biological: cerebro-spinal fluid — 1 ml of cerebro-spinal fluid

SUMMARY:
The study aims at identifying the type of B and CD4 T cell subsets with pathogenic properties in the different clinical forms of multiple sclerosis. This research might open new therapeutic approaches for the treatment of multiple sclerosis particularly progressive MS.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic autoimmune disease damaging the central nervous system (CNS). MS is categorized into several distinct forms according to clinical symptoms and medical examinations. Relapsing-remitting multiple sclerosis (RRMS) is characterized by attacks of worsening neurologic function, followed by partial or complete recovery periods. Patients can also present a gradual but steady progression of the disease (progressive forms). While several treatment options are currently available, no treatment completely stops the disease progression. Therefore, a deeper understanding regarding the mechanism of the disease development is essential to generate more efficient treatment strategies. CD4 T cells are known to be significantly involved in the formation of the CNS lesions characteristic of MS.The investigators hypothesize that different types of B and CD4 T cells play major roles in different forms of the disease. They will determine the phenotype and functions of the cells from the immune system particularly B and CD4 T cells present in the blood and cerebro-spinal fluid (CSF) of patients diagnosed with multiple sclerosis or presenting a clinically isolated syndrome.

The study will recruit 150 patients followed in Bordeaux University Hospital and diagnosed for clinically isolated syndrome (CIS) or multiple sclerosis (MS). Blood and CSF will be collected during a scheduled visit to study the properties of cells from the immune system in particular CD4 T cells in multiple sclerosis. Clinical and biological disease activity, treatment and outcomes will be studied in correlation with the properties of blood and CSF lymphocytes. No extra visit will be needed and the blood and CSF samples will be collected at the same times as those collected for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects ;
* Age ≥ 18 years;
* subjects with MS defined by 2010 revised McDonald criteria or presenting a clinical isolated syndrome;
* patients for which a blood draw and / or lumbar puncture to collect CSF is performed for diagnostic or therapeutic purpose;
* affiliated to an health insurance system;
* and who agree to participate in the study.

Exclusion Criteria:

* Pregnant or breastfeeding women,
* patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Functional and phenotypical characterization of the blood and CSF lymphocytes in MS and CIS patients. | At inclusion (day 0)

SECONDARY OUTCOMES:
Quantification of disease activity scores | At inclusion (day 0)
  Expanded Disability Status Scale (EDSS)
Quantification of disease activity scores | At inclusion (day 0)
  ambulation test
Number of lesions | At inclusion (day 0)
  evaluated by MRI
Size of lesions | At inclusion (day 0)
  evaluated by MRI
Localisation of lesions | At inclusion (day 0)
  evaluated by MRI
Types of lesions | At inclusion (day 0)
  evaluated by MRI
duration of the disease | At inclusion (day 0)
age at onset and progression | At inclusion (day 0)
number of relapses | At inclusion (day 0)
date of relapses | At inclusion (day 0)
Treatment | At inclusion (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie RUET, Prof, Principal Investigator — University Hospital, Bordeaux; Nathalie SCHMITT, PhD, Study Director — University of Bordeaux
Locations (1):
- CHU de Bordeaux - service de neurologie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No